CLINICAL TRIAL: NCT05642871
Title: DKI Combined With APT for Post-treatment Assessment of Ovarian Malignancies and Correlation With XRCC2 Gene
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianqian Qu (Other)
Responsible Party: Sponsor-Investigator, Qianqian Qu, Radiology, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: mr2022-10-01
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Malignant Tumor of the Ovary; XRCC2 Gene Mutation
MeSH Terms: conditions — Ovarian Neoplasms | interventions — APT

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — XRCC2
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Magnetic Resonance Multifunctional Imaging
  Interventions: Radiation: DKI and APT

INTERVENTIONS:
Radiation: DKI and APT — DKI and APT in patients with ovarian malignancy before and after treatment

SUMMARY:
Ovarian cancer is one of the common causes of cancer death in women worldwide. Despite the continuous development of diagnostic and treatment techniques, the survival rate of ovarian cancer patients has not improved significantly, and the important reason for the high mortality rate and poor prognosis is the lack of effective means to assess the effectiveness of treatment. The methods to monitor the effectiveness of ovarian cancer treatment and dynamic risk stratification by conventional imaging or single tumour marker levels are rather limited. In recent years, DKI and APT imaging have made some achievements in evaluating the post-treatment outcome of tumours, and the quantitative parameters of DKI combined with APT as a non-invasive biological marker are expected to be an effective way to address the limitations of assessing the treatment outcome by non-invasively detecting the changes in the signal of water protons and the diffusion information of non-normally distributed water molecules in the tumour tissue to observe the changes of protein and microstructure in the tumour cells. This project aims to collect patients who have come to our hospital for treatment. This project aims to collect patients with ovarian malignancies who come to our hospital and perform DKI, APT sequence and XRCC2 gene examination before and after treatment, and to statistically analyse the obtained parameters to assess the value of DKI combined with APT in monitoring the treatment effect of ovarian malignancies and the correlation with XRCC2 gene. This will help to promote individualised and precise treatment of ovarian cancer and improve prognosis.

ELIGIBILITY:
Inclusion Criteria:

No previous history of ovarian tumours or ovarian surgery; no concurrent other tumours, no history of oncology or treatment such as radiotherapy or chemotherapy; confirmed by pathological histology; receiving chemotherapy with a combination of platinum and purple shirt for at least 3 cycles; no contraindications to MRI

Exclusion Criteria:

Recurrent ovarian malignancy; too old, poor physical infrastructure; severe medical comorbidity; incomplete patient data collection; lost to follow-up

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with first diagnosis of ovarian malignancy; enrolled patients receive paclitaxel + cisplatin combination chemotherapy in 3-week cycles, with efficacy assessed every 3 cycles
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2023-01-31 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
DKI diffusion indicators and APT signal values | 2 Years
  MK MD SI

IPD SHARING:
Plan to Share IPD: Undecided